CLINICAL TRIAL: NCT01090687
Title: Role of 3D Tomography in Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: URMC-UMASS; 1R21CA134128-01A2 (NIH)
Record Dates: First submitted 2010-02-22; First posted 2010-03-22 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: breast cancer, CT scans, mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group I Microcalcifications: After classification as BI-RADS 4/5, approximately 75 to 100 subjects with primary findings based on microcalcifications will be recruited to have a breast CT scan.
  Interventions: Radiation: computed tomography (CT scan)
- Group II Soft tissue findings: After classification as BI-RADS 4/5, approximately 75 to 100 subjects with primary soft tissue findings, with or without associated microcalcifications, will be recruited to have a breast CT scan.
  Interventions: Device: computed tomography (CT scan)

INTERVENTIONS:
Radiation: computed tomography (CT scan) — Subjects will undergo cone beam breast CT scan
  Other Names: CT scan
  Groups: Group I Microcalcifications
Device: computed tomography (CT scan) — Subjects will undergo cone beam breast CT scan
  Other Names: CT scan
  Groups: Group II Soft tissue findings

SUMMARY:
The primary aim of this pilot study is to define the role of dedicated cone beam breast computed tomography in breast cancer imaging. This research is a prelude of a more comprehensive clinical trial that may follow.

ELIGIBILITY:
Inclusion Criteria:

* All women, age 40 or older, who are scheduled for biopsy after classification as BI-RADS 4/5 and have had a screening or diagnostic full-field digital mammography (FFDM) exam are eligible to participate, except for exclusions noted below.
* Able to provide informed consent.

Exclusion Criteria:

* Males
* Women less than 40 years old
* Pregnant women
* Lactating women
* Woman who have had bilateral mastectomies
* Women with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker
* Women who are unable to tolerate study constraints, frail or unable to cooperate
* Women with large breasts that cannot be accommodated within the field of view of the CT system
* Women who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to)

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkin's disease
* Women who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Women who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to)

  * Tuberculosis
  * Severe scoliosis

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, age 40 or older, who are scheduled for biopsy after classification as BI-RADS 4/5 and have had a screening or diagnostic full-field digital mammography (FFDM) exam, and who meet the inclusion criteria, are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Correlation between mammography and breast CT on lesion detection | 2 years
  There are two specific aims of this pilot study. One specific aim is to determine if the lesions that are detected by mammography and referred for biopsy, are visible with breast CT. The other specific aim is to determine if there is a correlation between CT numbers and malignancy, in particular for soft tissue (solid masses) abnormalities and to determine if image processing techniques improve correlation between CT numbers and malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Karellas, PhD, Principal Investigator — University of Massachusetts, Worcester; Stephen Glick, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Rochester Medical Center, Highland Breast Imaging Center, Rochester, New York, United States